CLINICAL TRIAL: NCT01289275
Title: Smoking Cessation in Hospitalized Smokers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Shu-Hong Zhu, Professor, University of California, San Diego
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 1U01CA159533-01 (NIH); 5U01CA159533 (NIH)
Record Dates: First submitted 2011-01-31; First posted 2011-02-03 (Estimated); Results first posted 2017-11-29 (Actual); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Smoking Cessation
Keywords: tobacco cessation; smoking cessation; telephone; self-help; smoking abstinence; tobacco use disorder; hospital; cardiopulmonary diseases; disparity
MeSH Terms: conditions — Smoking Cessation; Tobacco Use Cessation; Tobacco Use Disorder; Pulmonary Heart Disease | interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Telephone Counseling (Experimental): Up to 5 proactive counseling sessions
  Interventions: Behavioral: Telephone Counseling; Behavioral: Brief Hospital Counseling
- Nicotine Patches (Experimental): 8 weeks of nicotine patches
  Interventions: Drug: Nicotine Patches; Behavioral: Brief Hospital Counseling
- Telephone Counseling + Patches (Experimental): 5 proactive sessions, 8 weeks patches
  Interventions: Drug: Nicotine Patches; Behavioral: Telephone Counseling; Behavioral: Brief Hospital Counseling
- Brief hospital counseling (Active Comparator): brief in hospital counseling, no proactive sessions or patches
  Interventions: Behavioral: Brief Hospital Counseling

INTERVENTIONS:
Drug: Nicotine Patches — Subjects randomized into the patch condition will receive 8 weeks of nicotine patches at discharge. The kit will contain 4 weeks of 21mg patches, 2 weeks of 14mg, and 2 weeks of 7mg.
  Arms: Nicotine Patches; Telephone Counseling + Patches
Behavioral: Telephone Counseling — Up to 5 proactive counseling sessions from California Smokers' Helpline.
  Arms: Telephone Counseling; Telephone Counseling + Patches
Behavioral: Brief Hospital Counseling — All subjects receive bedside counseling either from Respiratory Therapists or nurses according to the hospital's particular practices.

SUMMARY:
When smokers are hospitalized they quit smoking, either voluntarily or involuntarily. Most of them, however, go back to smoking soon after discharge. This study will test an innovative approach which includes dispensing nicotine patches at discharge, providing proactive telephone counseling post discharge, or giving a combination of the two. The interventions are aimed at increasing the long term quit rate of these patients.

The specific aims of the study are to demonstrate the effects of two interventions, dispensing nicotine patches at discharge and providing proactive telephone counseling soon after discharge, on 12-month quit rates of hospitalized smokers in a 2 x 2 factorial design.

DETAILED DESCRIPTION:
Most smokers in the U.S. actually do quit smoking when hospitalized, either voluntarily or involuntarily because of hospital's nonsmoking policy. However, the majority of them return to smoking soon after their discharge from the hospital. A hospital stay, therefore, is a "teachable moment" for these patients, a good opportunity to encourage them to lead a smoke-free life after they are discharged. Research, however, has found that brief counseling provided to smokers while they are hospitalized has limited effect. The scientific data clearly show that smokers should be identified at the hospital, provided counseling, and given intensive interventions with follow up extended to 1 month post discharge. Providing such clinical services to these patients will reduce their chance of relapse to smoking and the rate of re-hospitalization. In practice though, hospitals have had difficulty providing even basic bedside counseling with a subgroup of patients, not to mention a much longer follow up post-discharge with all patients.

The proposed study aims to demonstrate that state quitlines can help bridge the gap between the recommendations from existing scientific data and the current practice by hospitals. Quitlines deliver counseling services by telephone. This is convenient for patients because they do not have to go anywhere in order to receive the counseling. Moreover, telephone counseling can be delivered proactively by the counselor.

The potential impact of this study is that if this model is proven effective in a rigorous study design, then it is likely that state quitlines across the U.S. will adopt it and start working with hospitals that are interested in using such as system. If the new JCAHO requirements get adopted, there will be a strong incentive for the hospitals to work with partners like the quitlines that can help provide follow up counseling.

With the proposed project the investigators intend to establish a practical model that lends itself to broader dissemination, while testing the effectiveness of the interventions with the rigor of a randomized design.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Smoke >=6 Cigarettes per day
* English or Spanish speaking
* Valid phone number
* Valid address
* Gave consent to participate in study and evaluation

Exclusion Criteria:

* Hospital stay of less than 24 hours
* Inability to communicate orally
* Hypersensitivity to nicotine
* Pregnant
* Hospitalized for psychiatric treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1270 (Actual)
Dates: Start 2011-08; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shu-Hong Zhu, Ph.D., Principal Investigator — UCSD
Locations (6):
- United States (6):
  - Scripps Mercy - Chula Vista, Chula Vista, California
  - Univeristy of California, Davis, Davis, California
  - UCSD - Thornton Hospital, La Jolla, California
  - Scripps Mercy - San Diego Campus, San Diego, California
  - UCSD Medical Center - Hillcrest, San Diego, California
  - University of California, San Diego: California Smokers' Helpline, San Diego, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cummins SE, Gamst AC, Brandstein K, Seymann GB, Klonoff-Cohen H, Kirby CA, Tong EK, Chaplin E, Tedeschi GJ, Zhu SH. Helping Hospitalized Smokers: A Factorial RCT of Nicotine Patches and Counseling. Am J Prev Med. 2016 Oct;51(4):578-86. doi: 10.1016/j.amepre.2016.06.021. PMID 27647058
- [Derived] Duffy SA, Cummins SE, Fellows JL, Harrington KF, Kirby C, Rogers E, Scheuermann TS, Tindle HA, Waltje AH; Consortium of Hospitals Advancing Research on Tobacco (CHART). Fidelity monitoring across the seven studies in the Consortium of Hospitals Advancing Research on Tobacco (CHART). Tob Induc Dis. 2015 Sep 3;13(1):29. doi: 10.1186/s12971-015-0056-5. eCollection 2015. PMID 26336372
- [Derived] Cummins S, Zhu SH, Gamst A, Kirby C, Brandstein K, Klonoff-Cohen H, Chaplin E, Morris T, Seymann G, Lee J. Nicotine patches and quitline counseling to help hospitalized smokers stay quit: study protocol for a randomized controlled trial. Trials. 2012 Aug 1;13:128. doi: 10.1186/1745-6215-13-128. PMID 22853197

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Smokers hospitalized at participating healthcare systems UCSD, Scripps, and UC Davis) between August 2011 and November 2013.
Pre-assignment Details: Inclusion criteria: adults, speak and read English or Spanish, smoked prior to hospitalization, cigarette consumption greater than 5 cigarettes per day.
Groups:
- Telephone Counseling: Telephone Counseling: Proactive. Counseling includes a 30-40 minute comprehensive pre-quit session plus up to 5 shorter follow-up calls (about 10 minutes) that are scheduled according to the probability of relapse. Counselors use a structured protocol so that there will be a record for each counseling call.
- Telephone Counseling and Nicotine Patches: Nicotine Patches: 8 weeks of nicotine patches at discharge.
  Telephone Counseling: Proactive. Counseling includes a 30-40 minute pre-quit session plus up to 5 shorter follow-up calls (about 10 minutes) that are scheduled according to the probability of relapse.
Period: Overall Study
Arm/Group | Telephone Counseling | Nicotine Patches | Telephone Counseling and Nicotine Patches | Brief Hospital Counseling
Started | 317 | 320 | 317 | 316
Completed | 317 | 320 | 317 | 316
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Telephone Counseling | Nicotine Patches | Telephone Counseling and Nicotine Patches | Brief Hospital Counseling | Total
Number analyzed (Participants) | 317 | 320 | 317 | 316 | 1270
Age, Continuous [Mean (Standard Deviation); unit: years] — years old at enrollment
  years | 48.2 (13.2) | 51.1 (13.5) | 49.1 (13.0) | 49.6 (13.0) | 49.9 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 136 | 134 | 144 | 136 | 550
  Male | 181 | 186 | 173 | 180 | 720
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 74 | 72 | 73 | 75 | 294
  Not Hispanic or Latino | 243 | 248 | 244 | 241 | 976
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 5 | 3 | 1 | 11
  Asian | 9 | 7 | 11 | 6 | 33
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 49 | 62 | 59 | 66 | 236
  White | 165 | 163 | 160 | 158 | 646
  More than one race | 15 | 8 | 8 | 15 | 46
  Unknown or Not Reported | 77 | 75 | 76 | 70 | 298
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 317 | 320 | 317 | 316 | 1270

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With 30-day Abstinence
Description: All participants will receive an assessment Interview 6-months after their initial contact with the Helpline. The interview will cover, as appropriate, tobacco use, use of quitting aids, pattern of quitting (including slips and relapse situations), and satisfaction with the services. The interview will be conducted over the telephone. Intention to treat analysis.
Time Frame: 6-months post enrollment
Population: all randomized subjects
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Telephone Counseling | Nicotine Patches | Telephone Counseling and Nicotine Patches | Brief Hospital Counseling
Number analyzed (Participants) | 317 | 320 | 317 | 316
percentage of participants | 18.0 [13.7 to 22.2] | 23.4 [18.8 to 28.1] | 22.1 [17.5 to 26.7] | 18.7 [14.4 to 23.0]

2. Secondary Outcome: Percentage of Smokers Making a 24-hour Quit Attempt
Time Frame: 6-months post enrollment
Population: all randomized subjects
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Telephone Counseling | Nicotine Patches | Telephone Counseling + Patches | Brief Hospital Counseling
Number analyzed (Participants) | 317 | 320 | 317 | 316
percentage of participants | 70.0 [63.8 to 76.3] | 78.9 [73.5 to 84.3] | 77.6 [72 to 83.2] | 69.7 [63.6 to 75.8]

3. Secondary Outcome: Self-reported Re-hospitalization
Time Frame: 6-months post enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Telephone Counseling | Nicotine Patches | Telephone Counseling + Patches | Brief Hospital Counseling
Number analyzed (Participants) | 317 | 320 | 317 | 316
Participants | 45 | 50 | 53 | 51

4. Secondary Outcome: 30-day Abstinence
Description: All participants will receive an assessment Interview 2-months after their initial contact with the Helpline. The interview will cover, as appropriate, tobacco use, use of quitting aids, pattern of quitting (including slips and relapse situations), and satisfaction with the services. The interview will be conducted over the telephone.
Time Frame: 2-months post enrollment
Population: all randomized subjects
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Telephone Counseling | Nicotine Patches | Telephone Counseling + Patches | Brief Hospital Counseling
Number analyzed (Participants) | 317 | 320 | 317 | 316
percentage of participants | 19.6 [15.2 to 23.9] | 22.5 [17.9 to 27.1] | 24.0 [19.3 to 28.7] | 18.4 [14.1 to 22.6]

ADVERSE EVENTS:
Time Frame: Data were collected over 7 months, ending with the 7 month post-enrollment evaluation.
Description: Rehospitalization was asked at the time of evaluation.
Arm/Group | Telephone Counseling | Nicotine Patches | Telephone Counseling and Nicotine Patches | Brief Hospital Counseling
All-Cause Mortality (participants affected / at risk) | 8/317 | 11/320 | 15/317 | 9/316
Serious Adverse Events (participants affected / at risk) | 69/317 | 77/320 | 76/317 | 88/316
Other Adverse Events (participants affected / at risk) | 0/317 | 0/320 | 0/317 | 0/316
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Telephone Counseling (N=317) | Nicotine Patches (N=320) | Telephone Counseling and Nicotine Patches (N=317) | Brief Hospital Counseling (N=316)
rehospitalization (General disorders) | 69 (69) | 77 (77) | 76 (76) | 88 (88) — rehospitalization with yes/no. The reason for rehospitalization was not established so we cannot designate the organ system

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No